CLINICAL TRIAL: NCT01461551
Title: Different Effects of Sevoflurane, Propofol and Combine of Sevoflurane and Propofol Maintained Anesthesia on Peripheral Blood Lymphocytes During Off-pump Coronary Artery Bypass Graft Surgery
Brief Title: Anesthesia and Lymphocytes Apoptosis
Acronym: OPCAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Li-Jie Jia, resident, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OPCAB
Record Dates: First submitted 2011-10-19; First posted 2011-10-28 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Anesthesia
Keywords: troponin I; creatine kinase mb; hospital days; lymphocyte apoptosis; intensive care unit days
MeSH Terms: interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sevoflurane (Experimental)
  Interventions: Drug: Sevoflurane
- Propofol (Experimental)
  Interventions: Drug: Propofol
- Combine of sevoflurane and propofol (Experimental)
  Interventions: Drug: combine of sevoflurane and propofol

INTERVENTIONS:
Drug: Sevoflurane — anesthesia was maintained with sevoflurane (end-tidal concentration 1.0-1.5 minimum alveolar concentration)
  Arms: Sevoflurane
Drug: Propofol — anesthesia was maintained with propofol (2-4 μg/ml via target-controlled infusion)
  Arms: Propofol
Drug: combine of sevoflurane and propofol — anesthesia was maintained with a combine of propofol (1 μg/ml via target-controlled infusion) and sevoflurane (end-tidal concentration 0.7-1.0 minimum alveolar concentration)
  Arms: Combine of sevoflurane and propofol

SUMMARY:
Most researches revealed that volatile anesthetic sevoflurane has a more marked cardioprotective effect against ischemia compared with intravenous agent propofol.However, propofol has been suggested to be more benefit for attenuation of surgery-induced immunosuppression.Thus, the aim of this study was to investigate under the specific OPCAB surgical stress, the influence of 3 established anesthetic techniques: sevoflurane, propofol and combine of sevoflurane and propofol maintained anesthesia on the apoptosis of circulating lymphocytes.

ELIGIBILITY:
Inclusion Criteria:

* male adults
* aged 18-80 yr
* undergoing elective OPCAB surgery containing left anterior descending artery bypass

Exclusion Criteria:

* a previous unusual response to any of the experimental anesthetics
* severe cardiac dysrhythmias or ejection fraction below 30%
* hemodynamic instability
* previous surgical coronary artery repair
* anemia, abnormal leukocytes or coagulopathy
* severe hypertension
* severe hepatic (albumin<30g,ascites), renal (serum creatinine greater than 2.0 mg/dl) or pulmonary (preoperative pulmonary function tests moderate-severe) dysfunctions
* concomitant surgical procedures and psychiatric disorders
* Insulin-dependent diabetics

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-10; Primary Completion 2012-02 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bu-Wei Yu, Ph.D., M.D., Study Director — Department of Anesthesiology, Ruijin Hospital, Shanghai Jiao tong University School of Medicine
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Jia L, Dong R, Zhang F, Wang W, Lu H, Luo Y, Xue Q, Yu B. Propofol Provides More Effective Protection for Circulating Lymphocytes Than Sevoflurane in Patients Undergoing Off-Pump Coronary Artery Bypass Graft Surgery. J Cardiothorac Vasc Anesth. 2015 Oct;29(5):1172-9. doi: 10.1053/j.jvca.2015.01.008. Epub 2015 Feb 19. PMID 26205644
- See also: Related Info — http://www.shsmu.edu.cn/
- See also: Related Info — http://www.sjtu.edu.cn/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment took place from October 9, 2011 to January 12, 2012 in Ruijin Hospital. A total of 149 patients scheduled to undergo elective OPCABG surgery were assessed for eligibility, with 105 patients enrolled and allocated randomly.
Pre-assignment Details: A total of 105 patients enrolled and allocated randomly. Five of these patients were excluded after enrollment (four due to changes in surgical schedules, and one due to severe hemodynamic instability during clamping of the coronary artery and requiring cardiopulmonary bypass).
Period: Overall Study
Arm/Group | Sevoflurane | Propofol | Combine of Sevoflurane and Propofol
Started | 35 | 35 | 35
Completed | 33 | 34 | 33
Not Completed | 2 | 1 | 2
Not completed — Physician Decision | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sevoflurane | Propofol | Combine of Sevoflurane and Propofol | Total
Number analyzed (Participants) | 33 | 34 | 33 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (8) | 62 (8) | 65 (9) | 63 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 33 | 100
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 33 | 34 | 33 | 100

OUTCOME MEASURES:

1. Primary Outcome: Lymphocyte Count
Description: Blood samples were obtained 24 h after the surgery for routine blood examination. This analysis was performed in the hospital laboratory using routine laboratory procedures.
Time Frame: 1 day after surgery
Measure: Mean (Standard Deviation); unit: cells/nanoliter
Arm/Group | Sevoflurane | Propofol | Combine of Sevoflurane and Propofol
Number analyzed (Participants) | 33 | 34 | 33
cells/nanoliter | 0.55 (0.25) | 0.73 (0.27) | 0.73 (0.31)

2. Secondary Outcome: Intensive Care Unit Staying Days
Time Frame: participants will stay in intensive care unit after surgery, an expected average of 2 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Sevoflurane | Propofol | Combine of Sevoflurane and Propofol
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/34 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes